CLINICAL TRIAL: NCT00022009
Title: Phase I/II Randomized Trial Comparing Two Treatment Schedules Of Gemcitabine In Poor Prognosis Status Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Gemcitabine Plus Supportive Care in Treating Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068683; CHNT-GEM; EU-20062
Record Dates: First submitted 2001-08-10; First posted 2003-06-12 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2002-10

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine

INTERVENTIONS:
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Treatment plus supportive care may improve quality of life in patients undergoing cancer treatment.

PURPOSE: Randomized phase II/III trial to compare the effect of different gemcitabine regimens plus supportive care on quality of life in patients who have locally advanced or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare quality of life, in terms of the degree of symptom palliation and improvements in performance status, of patients with locally advanced or metastatic poor prognosis non-small cell lung cancer treated with 2 schedules of gemcitabine combined with best supportive care.
* Compare the toxicity of these regimens in these patients.
* Compare the overall survival of patients treated with these regimens.
* Compare the response rate in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive gemcitabine IV over 30 minutes once a week for 3 weeks. Treatment continues every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive gemcitabine IV over 30 minutes once a week for 2 weeks. Treatment continues every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients on both arms also receive best supportive care. Additional courses of gemcitabine may be administered at the discretion of the investigator.

Quality of life is assessed at baseline and then after each course of chemotherapy.

Patients are followed every 2 months for survival.

PROJECTED ACCRUAL: A total of 174 patients (87 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven locally advanced or metastatic non-small cell lung cancer that is not amenable to curative surgery or radiotherapy
* No known CNS metastases
* No concurrent cord compression or superior vena cava syndrome requiring immediate radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 40-70%

Life expectancy:

* At least 4 weeks

Hematopoietic:

* WBC at least 3,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 10.0 g/dL

Hepatic:

* Bilirubin no greater than 3 times normal
* ALT and AST no greater than 3 times normal (5 times normal if liver metastasis present)

Renal:

* Creatinine no greater than 1.5 times normal

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 3 months after study
* No active infection
* No other concurrent serious, systemic disorder that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent systemic chemotherapy

Endocrine therapy:

* Concurrent steroids allowed

Radiotherapy:

* See Disease Characteristics
* Concurrent palliative radiotherapy allowed
* No concurrent curative radiotherapy

Surgery:

* See Disease Characteristics
* Concurrent palliative surgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07

CONTACTS AND LOCATIONS:
Overall Officials: Nick Thatcher, PhD, FRCP, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom